CLINICAL TRIAL: NCT01759667
Title: Diet-induced Thermogenesis After Roux-en-Y Gastric Bypass - A Prospective Study
Brief Title: DIT After RYGB - A Prospective Study
Acronym: DIT RYGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Leite Faria (Other)
Responsible Party: Sponsor-Investigator, Silvia Leite Faria, Nutritionist, Master of Science in Human Nutrition, Gastrocirurgia, Brazil
Organization: Gastrocirurgia, Brazil (Other)
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2012-12-14; First posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Obesity; Morbid Obesity; Bariatric Surgery
Keywords: Diet-induced Thermogenesis;; Respiratory Quotient;; Roux-en-Y Gastric Bypass;; Energy Expenditure.
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A standard mixed Meal (Experimental): The standard mixed meal was composed of a chicken salad sandwich and 200ml of coconut water, totalling 260 kcal, distributed among carbohydrates (62%), proteins (12%) and lipids (26%).
  Interventions: Other: A standard mixed Meal

INTERVENTIONS:
Other: A standard mixed Meal — All patients underwent an indirect calorimetry test, after a 12-h period of fasting from food and water, avoiding intake of alcohol or coffee, and avoiding physical exercise and cigarettes the day before the examination. To examine possible changes in the thermogenic effect of food, patients received a standard mixed meal (200 ml coconut water and a chicken salad sandwich using whole wheat bread). They then repeated the test 20 min and 60 min after eating to obtain a reading of the metabolic rate by considering DIT and the RQ in the postprandial period.

SUMMARY:
Bariatric surgery is the only satisfactory treatment for loss and weight maintenance in obese patients. This loss is a result of several factors that go beyond the simple anatomical abnormality of the gastrointestinal tract and may be the product of post-op energy expenditure changes. The respiratory quotient (RQ) and diet-induced thermogenesis (DIT) are important components of energy expenditure and possible changes in them can perform an important role in weight loss after Roux-en-Y Gastric Bypass (RYGB). Previously, we conducted a cross-sectional study where we measured the RQ and DIT in pre and post-op RYGB patients, which was published in the Surgery of Obesity and Related Diseases (SOARD) journal. The objective of this study is to perform a prospective analysis of these same variables (RQ and DIT), evaluating them in the same patients, when pre and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Pre-op: Body mass index (BMI) ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 with associated co-morbidities. Age > 18 years
* Post-op: Patients who underwent surgery ≥ 12 months by the Head Surgeon of the Gastrocirurgia de Brasilia Clinic;

Exclusion Criteria:

* Patients aged > 65 years. Severe heart and/or respiratory problems; Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Post-op DIT increase | 2 months
  A post-op increase in DIT is expected to be greater than in pre-op period and may be a positive predictor for weight loss during the post-op phase.

SECONDARY OUTCOMES:
Post-op RQ increase | 2 months
  A postprandial increase in RQ greater than that in the pre-op phase is expected showing improvement in carbohydrate metabolism after RYGB.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia L Faria, M.Science, Principal Investigator — Gastrocirurgia de Brasilia
Locations (1):
- Gastrocirurgia de Brasilia, Brasília, Federal District, Brazil